CLINICAL TRIAL: NCT06296433
Title: Extended Reality-Assisted Therapy for Chronic Pain Management: Can Immersive Virtual Reality Improve Range of Motion and Disability in Patients With Chronic Low Back Pain?
Brief Title: Extended Reality-Assisted Therapy for Chronic Pain Management
Acronym: XR-PAIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut d'Investigacions Biomèdiques August Pi i Sunyer (Other)
Responsible Party: Principal Investigator, Prof. Maria V. Sanchez-Vives, Professor, Institut d'Investigacions Biomèdiques August Pi i Sunyer
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCB_2023_1196
Record Dates: First submitted 2024-02-29; First posted 2024-03-06 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Chronic Pain; Low Back Pain
Keywords: virtual reality; embodiment; chronic pain; rehabilitation
MeSH Terms: conditions — Chronic Pain; Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR rehabilitation treatment (Experimental): Daily use of VR rehabilitation program independently at home for a period of 3 weeks. Each daily session is 20 minutes.
  Interventions: Other: VR rehabilitation
- VR control treatment (Placebo Comparator): Daily watching 2D video independently at home using VR headset for a period of 20 minutes.
  Interventions: Other: VR video application

INTERVENTIONS:
Other: VR rehabilitation — VR software application containing education, exergames, therapeutic exercises and relaxation sections.
  Arms: VR rehabilitation treatment
Other: VR video application — VR software application that plays 2D nature videos
  Arms: VR control treatment

SUMMARY:
The goal of this clinical trial is to test a home-based virtual reality rehabilitation application in patients with chronic low back pain. The main question it aims to answer are:

Is a prototype of a novel VR software application effective at reducing pain, improving daily function, improving range of motion, and reducing fear of movement in adult patients with chronic low back pain compared with a passive VR intervention? Participants in the treatment group will use the application daily for 20 minutes for a period of 3 weeks at home and unsupervised. Researchers will compare use of the VR application with a control group that watches 2D video to see if the treatment group have improved pain, disability, range of motion, and fear of movement.

DETAILED DESCRIPTION:
This is a two-arm randomized parallel controlled trial designed to test a prototype of a VR software application that the investigators have developed for patients with chronic low back pain. The app contains (1) educational messages delivered by a virtual therapist, (2) gamified exercises in which the patient has to move to reach goals or avoid objects, (3) therapeutic exercises, in which patients perform difficult or feared movements, (4) relaxation/mindfulness. There will be two groups consisting of adult patients of both sexes with persistent low back pain. Patients (n = 100) will be randomly assigned to either an interventional VR treatment (n = 50) or a control treatment (n = 50).

Patients in the VR intervention group will use the VR software application daily for a 20-minute training program. In the virtual reality application, they will be embodied into an avatar through congruent visuotactile and visuomotor stimulation (observed in first person) and will perform gamified movements and exercises for 15-20 minutes. These exercises will increase in difficulty for 3 weeks and will include educational and relaxation components. The control treatment will consist of a passive VR intervention in which the patient watches a TV show on a 2D screen but while wearing the virtual reality headset. They will be able to choose from three popular TV series with short episodes (20 minutes). The investigators will use validated outcome measures to assess changes in pain and function. These will be measured at baseline, after treatment (3 weeks), and at 1 month follow-up for both the treatment group and the control group. Both groups will be advised to continue their normal daily activities and routines, with no restrictions on activity or exercise, in addition to VR treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 of either sex
* Diagnosis of chronic low back pain of >12 weeks, with or without associated somatic referred leg pain
* Average pain intensity over the previous month ≤7/10 and ≥ 2/10)

Exclusion Criteria:

* Spondylolysis, fracture, cauda equina syndrome, active spinal infection
* Acute radiculopathy or compromised nerve root
* Recent spinal surgery (<12 months) or lower limb surgery (<3 months)
* Major depressive symptoms as indicated by the Patient Health Questionnaire-2 depression screen score of 4 or more.
* Current or prior diagnosis of epilepsy, seizure disorder, dementia, migraines, balance disorder, or other neurological diseases that may prevent the use of virtual reality or adverse effects.
* Cardiopulmonary or pulmonary disorder with contraindication to physical exercise
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Brief Pain Inventory | Baseline, 4 weeks, 8 weeks
  Allows patients to rate the severity of their pain and the degree to which their pain interferes with common dimensions of feeling and function. Minimum score 0, maximum score 70, higher score = worse outcome.

SECONDARY OUTCOMES:
Roland-Morris Disability Questionnaire | Baseline, 4 weeks, 8 weeks
  The Roland-Morris Disability Questionnaire is a self-reported measure consisting of 24 yes/no questions designed to assess functional disability related to back pain, with higher scores indicating greater disability. Minimum score 0, maximum score 24.
Short-Form 12 | Baseline, 4 weeks, 8 weeks
  The Short-Form-12 is a widely used, short-form health survey consisting of 12 questions that assess physical and mental health functioning, providing a concise measure of overall health status. Scores above 50 represent better than average quality of life, below 50 represents worse than average quality of life.
Patient Global Impression of Change | Baseline, 4 weeks, 8 weeks
  The Patient Global Impression of Change is a self-reported assessment used to measure an individual's perceived change in health status or symptoms over time, typically ranging from "very much worse" to "very much improved." Minimum score 1, maximum score 7. Higher score indicated greater improvement in patient's condition (better outcome)
Pain Catastrophization Scale | Baseline, 4 weeks, 8 weeks
  a self-report measure consisting of two subscales, assessing beliefs about how physical activity and work-related activities may exacerbate pain and lead to avoidance behaviors in individuals with low back pain. Minimum score 0, maximum score 52. Higher score indicates worse outcome.

OTHER OUTCOMES:
Spinal Range of motion | Baseline, 4 weeks, 8 weeks
  Video analysis will be used to measure spinal range of motion for flexion, extension and side flexion.
Adherence to treatment | 4 weeks
  Measured automatically in the VR headset
Embodiment | 4 weeks
  Self report questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Maria V Sanchez-Vives, Principal Investigator — Institut d'Investigacions Biomèdiques August Pi i Sunyer
Locations (1):
- IDIBAPS, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Study data will be made available on request from the study authors
Supporting Information: CSR
Time Frame: No time limit. Data will be made available on completion of the trial.
Access Criteria: Email request directly from Principle Investigator, Prof. Maria Sanchez-Vives (msanche3@recerca.clinic.cat)